CLINICAL TRIAL: NCT06370377
Title: Critical and Medical-Surgical Nurses' Adherence to Professional Nursing Code of Ethics and Quality of Nursing Care Satisfaction
Brief Title: Nurses' Adherence to Professional Nursing Code of Ethics and Quality of Nursing Care Satisfaction
Status: Completed | Type: Observational
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Other Study IDs: 0305899
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Professional Role; Nurse's Role; Ethics, Narrative; Satisfaction, Patient
MeSH Terms: conditions — Narration; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: the Egyptian code of ethical practice — Nurses' adherence to the Egyptian code of ethical practice

SUMMARY:
Nursing code of ethics is an essential part of nursing professional practice. Nurses' adherence to a code of ethics is an important pillar of improving their performance, providing good nursing care and achieving patient satisfaction.

DETAILED DESCRIPTION:
Nursing code of ethics is an essential part of nursing professional practice. Nurses' adherence to a code of ethics is an important pillar of improving their performance, providing good nursing care and achieving patient satisfaction.This study aimed to examine relationship between nurses' adherence to an Egyptian professional nursing code of ethical practice and patient satisfaction with quality of nursing care in critical and medical-surgical care units.

ELIGIBILITY:
Inclusion Criteria:

* Nurses

  * willing to participate in the study
  * work in surgical intensive and critical care units
  * Sign a consent
* Patients

  * Alert, conscious and educated patients
  * More than 18 years old

Exclusion Criteria:

* Nurses

  * Work in outpatient units and other units
  * Did not sign a consent
* Patients

  * Unaware or could not communicate
  * less than 18 years old

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Nurses: A convenience sampling was carried out on 400 nurses; 200 nurses in critical care units and 200 nurses in medical-surgical care units.400 alert, conscious and educated patients
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure source of nurses' knowledge about Egyptian code of ethics | one month
  source of nurses' knowledge about Egyptian code of ethics as assessed using a binary scale of yes=1 and no =0.
Observational checklist to measure | one month
  nurses' adherence to an Egyptian professional nursing code of ethical practice as assessed using three ranking scales (never practice (0 points) or sometimes practice (0.5 points) and always practice (1 point).
Questionnaire to measure patient satisfaction with the quality of nursing care | one month
  Patient satisfaction with quality of nursing care as assessed using five Likert scales ranging from 1 = poor and 5 = excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt; Safaa M. El-Shanawany, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Maha Ghanem, Ph.D, Study Chair — Forensic Medicine and Clinical Toxicology, Faculty of Medicine, Alexandria University, Egypt; Hanaa Abbass, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University , Egypt; Maysa Elbiaa, Ph.D, Principal Investigator — Faculty of Nursing, Matrouh University , Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No